CLINICAL TRIAL: NCT07078526
Title: Comparison of the Effectiveness of the Otago Exercise Program (Oep) and Neuromuscular Exercises on Pain, Functional Status, Postural Control, and Balance in Patients With Knee Osteoarthritis
Brief Title: Comparative Effectiveness of Otago and Neuromuscular Exercise Programs in Knee Osteoarthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0163
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Knee Osteoarthritis
Keywords: Otago Exercise Program; Neuromuscular Exercises; Knee Osteoarthritis; Pain Management; Functional Status; Postural Control; Balance
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a parallel manner to either the Otago Exercise Program group or the neuromuscular exercise group, receiving their assigned intervention concurrently over six weeks.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Exercise Program (Experimental): Participants in this arm will receive the Otago Exercise Program (OEP) consisting of 17 structured exercises (5 strengthening and 12 balance/proprioception exercises). Each session includes warm-up and cool-down, and lasts approximately 40 minutes. Sessions will be supervised twice weekly for a total duration of six weeks, in addition to standard physiotherapy (hot pack and gentle stretching).
  Interventions: Other: Otago Exercise Program
- Neuromuscular Exercise (Active Comparator): Participants in this arm will receive a structured neuromuscular exercise protocol including functional, proprioceptive, and balance exercises such as side stepping, high knees march, pelvic lifts, bridging with marching, lateral leg step, sit to stand, single leg clock reach, and single leg stand. Each session includes warm-up and cool-down, lasts approximately 40 minutes, and will be supervised twice weekly for six weeks, alongside standard physiotherapy (hot pack and gentle stretching).
  Interventions: Other: Neuromuscular Exercise

INTERVENTIONS:
Other: Otago Exercise Program — The Otago Exercise Program is a structured, progressive exercise regimen focusing on lower limb strengthening and balance retraining. It is performed twice weekly for six weeks under physiotherapist supervision, complementing standard physiotherapy care.
  Other Names: OEP
  Arms: Otago Exercise Program
Other: Neuromuscular Exercise — The neuromuscular exercise intervention involves functional, proprioceptive, and balance exercises delivered twice weekly for six weeks under supervision, in addition to standard physiotherapy care.
  Other Names: NME
  Arms: Neuromuscular Exercise

SUMMARY:
This randomized controlled trial aims to compare the effects of the Otago Exercise Program (OEP) and neuromuscular exercises on pain, functional status, postural control, and balance in patients with knee osteoarthritis (KOA). A total of 58 participants with X-ray confirmed Grade 2-3 KOA will be enrolled from clinical centers in Lahore, Pakistan. Eligible participants will be randomly assigned to either the OEP group or the neuromuscular exercise group. Both groups will receive standardized physiotherapy alongside their respective interventions twice weekly for six weeks. Outcomes including pain (NPRS), functional status (WOMAC), dynamic mobility (TUG), and postural control (mCTSIB) will be measured at baseline, week 3, and week 6. Data will be analyzed to determine which intervention provides greater improvements in pain reduction, functional capacity, mobility, and balance. This study is expected to inform clinical practice by identifying a more effective exercise approach for managing KOA symptoms and enhancing patients' quality of life.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a highly prevalent degenerative joint disease that significantly impairs mobility, functional capacity, and balance, often resulting in increased fall risk and reduced quality of life. Exercise-based interventions are widely recognized as key components of conservative management for KOA, yet comparative evidence for specific programs remains limited.

This randomized controlled trial is designed to compare the effectiveness of the Otago Exercise Program (OEP) and neuromuscular exercises in managing pain, improving functional status, enhancing postural control, and restoring balance in patients with Grade 2-3 knee osteoarthritis.

Eligible participants aged 45-65 years, with confirmed KOA and fulfilling inclusion criteria, will be recruited from multiple clinical centers in Lahore, Pakistan. After providing informed consent, participants will be randomized into two groups using computer-generated allocation with concealed envelopes.

Group A (OEP group) will receive the Otago Exercise Program, which consists of 17 structured exercises targeting lower limb strength and balance. Each session will include a warm-up, exercise circuit, and cool-down, conducted twice per week for six weeks under supervision.

Group B (neuromuscular group) will perform a series of neuromuscular exercises focused on functional, proprioceptive, and balance training. This protocol, also including warm-up and cool-down, will match the frequency and duration of the OEP group.

Both groups will receive standardized physiotherapy, including pain-relief modalities and gentle stretching exercises. Outcome measures, Numeric Pain Rating Scale (NPRS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Timed Up and Go (TUG), and Modified Clinical Test of Sensory Interaction in Balance (mCTSIB), will be collected at baseline, 3 weeks, and 6 weeks by an independent blinded assessor.

Data will be analyzed using appropriate parametric and non-parametric tests to evaluate within-group and between-group differences over time. It is hypothesized that both exercise interventions will yield significant improvements in pain and functional measures, but the Otago Exercise Program may offer superior benefits in balance and mobility performance.

Findings from this study are expected to guide clinicians in selecting effective exercise regimens to optimize rehabilitation outcomes and reduce the burden of knee osteoarthritis in the community.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 45 to 65 years
* X-ray confirmed Grade 2-3 knee osteoarthritis (Kellgren-Lawrence scale)
* NPRS pain score between 3 and 8
* TUG score ≥ 14 seconds
* Able and willing to participate in twice-weekly sessions for six weeks
* Signed informed consent

Exclusion Criteria:

* History of heart attack or stroke within the past year
* Knee or hip surgery within the past 6 months
* Resting systolic blood pressure >160 mmHg or <100 mmHg
* Resting diastolic blood pressure >100 mmHg or <60 mmHg
* Neurological disorders affecting balance
* Current participation in another exercise program
* Recent fractures, cancer, or vascular diseases

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | Baseline, Week 3, Week 6
  Pain intensity will be assessed using the Numeric Pain Rating Scale (NPRS), a validated 0-10 scale where higher scores indicate greater pain. Change from baseline to 6 weeks will be analyzed.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, Week 3, Week 6
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) will be used to measure pain, stiffness, and physical function in patients with knee osteoarthritis.
Timed Up and Go (TUG) | Baseline, Week 3, Week 6
  The Timed Up and Go (TUG) test will measure functional mobility by recording the time taken to stand up, walk 3 meters, return, and sit down.
Modified Clinical Test of Sensory Interaction in Balance (mCTSIB) | Baseline, Week 3, Week 6
  The Modified Clinical Test of Sensory Interaction in Balance (mCTSIB) will assess postural control by measuring sway under different sensory conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Mahnoor Butt, MSc OMPT, Principal Investigator — Riphah International University; Amna Zia, Phd Scholar, Principal Investigator — Mayo Hospital/ Riphah International University
Locations (1):
- Kulsoom Sultan Medical centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] .KATRE KA, PUSHPARAJ V, PAUL J. Effect of Otago Exercise Program (OEP) and Strength Training Program (STP) on leg strength and risk of fall among bilateral knee osteoarthritis patients. IJMAES. 2019;5(1):536-51.
- [Background] Tauqeer S, Shakeel H, Ikram A, Kafeel F, ul Ain N, Farooq N. Frequency of Grade (III) Knee Osteoarthritis (OA) Among Women in Lahore Pakistan: Grade (III) Knee Osteoarthritis (OA) Among Women. Pakistan BioMedical Journal. 2021;4(2):258-62.
- [Background] Rao RDM, Methe AD, Patil H, Prabhakar R. Effect of Otago exercise versus dual task net step exercise on balance and functional mobility in community dwelling elderly person with knee osteoarthritis-a randomised control trial. International Journal of Health Sciences and Research. 2021;11:179-87
- [Background] Malik FB, Memon AG, Shah S, Latif D, Afzal MF, Memon SA. PREVALENCE OF KNEE OSTEOARTHRITIS AND QUALITY OF LIFE AMONG MIDDLE AGED ADULTS OF PAKISTAN: soi: 21-2017/re-trjvol06iss01p280. The Rehabilitation Journal. 2022;6(01):280-3
- [Background] National Library of Medicine (U.S.). Exercise for osteoarthritis of the knee (NCT06329128). ClinicalTrials.gov. 2024. Available from: https://clinicaltrials.gov/ct2/show/NCT0632912
- [Background] Yang Y, Wang K, Liu H, Qu J, Wang Y, Chen P, Zhang T, Luo J. The impact of Otago exercise programme on the prevention of falls in older adult: A systematic review. Front Public Health. 2022 Oct 20;10:953593. doi: 10.3389/fpubh.2022.953593. eCollection 2022. PMID 36339194